CLINICAL TRIAL: NCT05658835
Title: Interest of Molecular Analysis of Cerebral Thrombi in Determining the Prognosis and Etiology of Cerebral Infarction
Acronym: MATISSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM22_0231; ID-RCB (Other: 2022-A01860-43)
Record Dates: First submitted 2022-12-08; First posted 2022-12-21 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-07

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; thrombi; metabolites
MeSH Terms: conditions — Ischemic Stroke; Thrombosis | interventions — Blood Coagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient suffering from ischemic stroke
  Interventions: Other: Thrombi and blood analyses

INTERVENTIONS:
Other: Thrombi and blood analyses — Thrombi and blood will be collected during thrombectomy

SUMMARY:
The MATISSE (Molecular Analysis of Thrombus for Ischemic Stroke prognosis and Etiology) project evaluates the hypothesis that the molecular composition of cerebral thrombus in metabolites, lipids, and proteins conditions the clinical prognosis at 3 months of the infarction and informs on its etiological subtype

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older;
* Patient with a cerebral infarction documented by brain imaging who received endovascular treatment by mechanical thrombectomy;
* Patient for whom it was possible to collect cerebral thrombus for LC-MS analysis during mechanical thrombectomy:
* Patient who was informed of the study and formulated a non-opposition to participation. If not, patient for whom a relative was informed and formulated a non-opposition.

Exclusion Criteria:

* Patient with a cerebral infarction documented by cerebral imaging, having benefited from an endovascular treatment with mechanical thrombectomy that did not allow the extraction of a cerebral thrombus.
* Protected persons (articles L1121-5, L1121-6 and L121-8 of the Public Health Code): pregnant or breast-feeding women, persons deprived of liberty, under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from ischemic stroke
Sampling Method: Probability Sample
Enrollment: 311 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-11-07 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Determination and validation of molecular signatures, obtained by LC-MS analysis of cerebral thrombi, predictive of the excellent clinical prognosis | 3 months after the cerebral infarction
  Rankin score (0 to 6, 6 meaning worse outcome)

SECONDARY OUTCOMES:
Determination and validation of molecular signatures, obtained by LC-MS analysis | 7 days after the cerebral infarction
  ASCOD (atherosclerosis, small vessel disease (SVD), cardioembolism, other and dissection) description (0 to 9, 9 meaning insufficient assessment to determine the presence or absence of the disease)
Determination and validation of molecular signatures, obtained by LC-MS analysis | 3 months after the cerebral infarction
  ASCOD (atherosclerosis, small vessel disease (SVD), cardioembolism, other and dissection) description (0 to 9, 9 meaning insufficient assessment to determine the presence or absence of the disease)
Severe intracranial hemorrhage | 3 months after the cerebral infarction
  Heildeberg classification (0 to 3d, 3d meaning subdural hemorrhage)
Recovery of autonomy in walking | 3 months after the cerebral infarction
  Parker score (0 to 9, 9 meaning better outcome)
Recovery of autonomy in walking | 7 days after the cerebral infarction
  Parker score (0 to 9, 9 meaning better outcome)
Early Neurological Deterioration | 24 hours after recanalization treatment
  Worsening of at least 4 points in the NIHSS (National Institutes of Health Stroke Scale) score (0 meaning better outcome, 0 to 42)
Use of thrombolytic therapy in the acute phase | Before thrombectomy
  Quantification of thrombolytic therapy
Determination of molecular signatures predictive on successful recanalization after mechanical thrombectomy | Right after the thrombectomy
  Score mTICI (modified Thrombolysis In Cerebral Infarction, 0 to 3, 0 meaning worst outcome)
Positive infarct growth after successful recanalization | Between 24 and 48h after the thrombectomy
  Quantification of infarctus volume by MRI
Death | 3 months after cerebral infarction
  Death of the patient
Patient exposure to peak outdoor air pollution | 96 hours before cerebral infarction
  Quantification of peak outdoor air pollution (identification of the location of the patient and the polluants observed in the areas)

CONTACTS AND LOCATIONS:
Overall Officials: François Crémieux, Study Director — AP-HM
Locations (4):
- France (4):
  - CHU Martinique, Fort-de-France
  - Stroke Center, Marseille
  - CHU Guadeloupe, Pointe à Pitre
  - CHU La Réunion, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No